CLINICAL TRIAL: NCT03306290
Title: An Evaluation of Serum Concentration of CEFOxitin Used for Antibiotic Prophylaxis in Severely and Morbidly Obese Patients Undergoing BARiatric Surgery (CEFOBAR)
Brief Title: Serum Concentration of CEFOxitin Used for Antibiotic Prophylaxis in Obese Patients Undergoing BARiatric Surgery
Acronym: CEFOBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A01285-48
Record Dates: First submitted 2017-08-28; First posted 2017-10-11 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Obese; Antibiotic Prophylaxis; Bariatric Surgery Candidate
Keywords: Obese; Bariatric surgery; Antibiotic prophylaxis; Cefoxitin
MeSH Terms: conditions — Obesity | interventions — Drug Dosage Calculations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bariatric surgery candidate (Other): Patients included in this study belong to this arm and put up with intervention "Serum dosage of antibiotic prophylaxis CEFOXITIN"
  Interventions: Drug: Serum dosage of antibiotic prophylaxis CEFOXITIN

INTERVENTIONS:
Drug: Serum dosage of antibiotic prophylaxis CEFOXITIN — Three blood samples will be collected. These samples are specific for the research, and will be performed on the forearm opposite to the one used for Cefoxitin infusion.
  1. Blood sample at the start of surgery (t0): at the end of the Cefoxitin infusion (~30 min), 1 tube (5 ml) of blood will be withdrawn
  2. Blood sample at half way surgery (t1): 1 tube (5 ml) of blood will be withdrawn (if applicable)
  3. Blood sample at skin closure (t2): 1 tube (5 ml) of blood will be withdrawn
  Other Names: Drug dosage

SUMMARY:
Obesity is a pandemic problem in modern societies. Bariatric surgery (gastric by-pass and sleeve gastrectomy) has emerged as an efficient treatment to reduce morbidity and mortality related to obesity. Obesity and bariatric surgery are known to be risk factors of surgical site infections (SSI). The occurrence of SSI increases health cost and the duration of hospitalization. However, an appropriate antibiotic prophylaxis has been shown to reduce SSI. As recommended by several national societies, the antibiotic prophylaxis dose should be increased in the severely obese population. However, this recommendation lies on a low level of evidence. Besides, great disparities regarding obese patient antibiotic prophylaxis exist between countries and adequate doses are still not clearly defined. In France, for instance, the intravenous second generation cephalosporin CEFOXITIN is used for antibiotic prophylaxis in bariatric surgery at the initial loading dose of 4g (2-fold that of non-obese population) at the beginning of surgery.

Obese patients have increased risk of under-dosage due to modification of their pharmacokinetics (fat/lean mass, distribution volume, renal clearance, etc.). Only few studies, all investigating a low amount of patients, evaluated the appropriateness of intraoperative antibiotic prophylaxis dosage of different betalactam and cephalosporin in the obese population. This population was more likely to be under-dosed.

The aim of this study is to analyse the appropriateness of the reference dose of intravenous Cefoxitin used as antibiotic prophylaxis in severely obese patients undergoing bariatric surgery. This will be a 2-year prospective monocentric study held in the University Hospital of Nancy, France. A large group of obese patients (~300) will be included. Serial serum concentration measurements of Cefoxitin will be performed before, during, and at skin closure of the bariatric surgery. This study will give insights in pharmacokinetics of the antibiotic prophylaxis in the obese population and will help to determine the initial dosage and the optimal method for antibiotic prophylaxis administration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years-old,
* Severely obese patient with a BMI ≥ 35 kg.m-2,
* Scheduled bariatric surgery: gastric by-pass or sleeve gastrectomy,
* Affiliated to social security,
* The patient is able to consent to clinical research and has received all information on the study design/protocol,
* Signed/written informed consent

Exclusion Criteria:

* Refuse to consent to the study or the patient is unable to consent,
* Allergy/Anaphylaxis to beta-lactam (ß-lactam) antibiotics either proven or suspected,
* Pregnancy,
* Persons deprived of their liberty by judicial or administrative decision,
* Urgent or emergent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Serum concentration of Cefoxitin at the beginning and end of the surgery with one extra measurement at halfway surgery | baseline
  Blood samples will be put at low temperature for transportation and then analysed by chromatographic method

SECONDARY OUTCOMES:
Identification of factors that may be associated with the risk of under-dosage | baseline
  effect of creatinine clearance on cefoxitine concentration
Identification of factors that may be associated with the risk of under-dosage | baseline
  effect of age of the patient on cefoxitine concentration
Identification of factors that may be associated with the risk of under-dosage | baseline
  effect of lenght of surgery on cefoxitine concentration
Identification of factors that may be associated with the risk of under-dosage | baseline
  effect of type of surgery on cefoxitine concentration
Pharmacokinetic parameters: drug clearance | baseline
  These parameters will be calculated according to the initial concentration (C0) and the final concentration (C2) measured at t0 and t2 respectively. A corrective factor will be applied according to the halfway surgery serum concentration of Cefoxitin.
  o Clearance: Cl=k x Vd
Pharmacokinetic parameter: volume of distribution | baseline
  This parameter will be calculated according to the initial concentration (C0) and the final concentration (C2) measured at t0 and t2 respectively. A corrective factor will be applied according to the halfway surgery serum concentration of Cefoxitin.
  o Volume of distribution: D0/C0
Pharmacokinetic parameter: half-life | baseline
  This parameter will be calculated according to the initial concentration (C0) and the final concentration (C2) measured at t0 and t2 respectively. A corrective factor will be applied according to the halfway surgery serum concentration of Cefoxitin.
  o Half-life: t1/2=ln2/k
Pharmacokinetic parameter: area under curve, | baseline
  This parameter will be calculated according to the initial concentration (C0) and the final concentration (C2) measured at t0 and t2 respectively. A corrective factor will be applied according to the halfway surgery serum concentration of Cefoxitin.
  o Area under curve: AUC=C0/k
Pharmacokinetic parameter: elimination rate | baseline
  This parameter will be calculated according to the initial concentration (C0) and the final concentration (C2) measured at t0 and t2 respectively. A corrective factor will be applied according to the halfway surgery serum concentration of Cefoxitin.
  o Elimination rate: k=(LnC0-LnC2)/(t2-t0)
Incidence of superficial incisional surgical site infection (SSI) at 30 days | up to 30 days after surgery
  o Superficial incisional SSI: at 30 days defined by:
  Date of event for infection occurs within 30 days after any operative procedure AND involves only skin and subcutaneous tissue of the incision AND the patient has at least one of the following:
  1. purulent drainage from the superficial incision,
  2. organisms identified from an aseptically-obtained specimen,
  3. from the superficial incision or subcutaneous tissue by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment (e.g., not Active Surveillance Culture/Testing (ASC/AST),
  4. superficial incision that is deliberately opened by a surgeon, attending physician or other designee and culture or non-culture based testing is not performed AND patient has at least one of the following signs or symptoms: pain or tenderness;localized swelling; erythema; or heat,
  5. diagnosis of a superficial incisional SSI by the surgeon or attending physician or other designee.
Incidence of deep incisional surgical site infection (SSI) at 30 days | up to 30 days after surgery
  Deep incisional SSI at 30 days defined by:
  date of event for infection occurs within 30 days after the operative procedure AND involves deep soft tissues of the incision (e.g., fascial and muscle layers) AND patient has at least one of the following:
  1. purulent drainage from the deep incision,
  2. a deep incision that spontaneously dehisces, or is deliberately opened or aspirated by a surgeon, attending physician or other designee and organism is identified by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment (e.g., not Active Surveillance Culture/Testing (ASC/AST) or culture or non-culture based microbiologic testing method is not performed AND patient has at least one of the following signs or symptoms: fever (>38°C); localized pain or tenderness.
  3. an abscess or other evidence of infection involving the deep incision that is detected on gross anatomical or histopathologic exam, or imaging test.
Incidence of organ/space surgical site infection (SSI) at 30 days | up to 30 days after surgery
  Organ/Space SSI at 30 days defined by:
  Date of event for infection occurs within 30 after the operative procedure AND infection involves any part of the body deeper than the fascial/muscle layers, that is opened or manipulated during the operative procedure AND patient has at least one of the following:
  1. purulent drainage from a drain that is placed into the organ/space
  2. organisms are identified from an fluid or tissue in the organ/space by a culture or non-culture based microbiologic testing method
  3. an abscess or other evidence of infection involving the organ/space that is detected on gross anatomical or histopathologic exam, or imaging test evidence suggestive of infection AND meets at least one criterion for a specific organ/space infection site listed: intraabdominal infection, not specified elsewhere including gallbladder, bile ducts, liver, spleen, pancreas, peritoneum, subphrenic or subdiaphragmatic space

CONTACTS AND LOCATIONS:
Overall Officials: El Mehdi SIAGHY, Study Director — Central Hospital, Nancy, France
Locations (1):
- Central Hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novy E, Liu X, Hernandez-Mitre MP, Belveyre T, Scala-Bertola J, Roberts JA, Parker SL. Population pharmacokinetics of prophylactic cefoxitin in elective bariatric surgery patients: a prospective monocentric study. Anaesth Crit Care Pain Med. 2024 Jun;43(3):101376. doi: 10.1016/j.accpm.2024.101376. Epub 2024 Mar 15. PMID 38494157